CLINICAL TRIAL: NCT01259193
Title: Phase II Study of Sorafenib and Zoledronic Acid in Advanced HCC
Brief Title: Clinical Study of Sorafenib and Zoledronic Acid to Treat Advanced HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Ren Zhenggang/Professor Sun Huichuan/Professor, Shanghai Zhongshan Hospital,China
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRFB-021; LCI-10-10-20
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2010-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Sorafenib; Zoledronic Acid; toxic reaction
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib and Zoledronic Acid (Experimental)
  Interventions: Drug: Sorafenib and Zoledronic Acid

INTERVENTIONS:
Drug: Sorafenib and Zoledronic Acid — Sorafenib ,tablet,400mg Bid ,until patient can not tolerance Zoledronic Acid ,powder for injection,4mg per 3 week for 1 year

SUMMARY:
Sorafenib ,an oral multikinase inhibitor targeting several tyrosine-kinase receptors with antiangiogenesis and antiproliferation of HCC, is the first approved target therapy for HCC.

Zoledronic acid is used for treatment of bone metastasis of diverse malignant cancer. Emerging data suggest that zoledronic acid may also exhibit anticancer properties.

The objectives of the study is to evaluate the safety of Sorafenib combined with Zoledronic Acid and to evaluate overall survival and time to progression.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Hepatocellular carcinoma confirmed with pathology or identified with radiological images with typical features
* patient with unresectable primary hepatocellular carcinoma
* Child-Pugh Class A or B, score ≤ 7
* ECOG score 0-2
* Expected survival time not less than 12 weeks
* At least one tumor nodule with one uni-dimension of ≥ 1 cm
* Peripheral platelet of or more than 50×10(9)/L
* Peripheral hemoglobin of or more than 85g/L
* Peripheral albumen of or more than 28g/L
* Total bilirubin ≤3.0mg/dl
* ALT and AST ≤ 5.0 x the upper limit of normal
* Serum amylase ≤ 1.5x the upper limit of normal
* Serum creatinine ≤ 1.5x upper limit of normal
* PT-INR<2.3 or PT prolong no more than 4s of normal

Exclusion Criteria:

* Congestive heart failure > NYHA class 2
* History of active coronary disease( except myocardial infarction more than 6 months ago)
* Receive anti-arrhythmia treatment(except β-receptor blocker,calcium channel blocker and digoxin)
* uncontrollable hypertension
* Active clinically serious infections (> 2 NCI-CTC Version 3.0)
* History of HIV infection
* Inclined to hemorrhage or active hemorrhage with 1 month
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in this study
* Pregnant or breast-feeding.Women of childbearing potential must have a negative pregnancy test performed within 7 days prior to enrolling in this portion of the study
* Known or suspected allergy to any agent given in association with this trial
* Concomitant anti-cancer therapy (except immunotherapy and Chinese traditional treatment)
* Surgical operation within 4 weeks prior to enrolling in this portion of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
numbers of adverse events | 1 year
  to evaluate the toxicity of sorafenib in combination with zoledronic acid

SECONDARY OUTCOMES:
Overall survival (OS), time to progression (TTP) | 1 year
  to evaluate the efficacy of sorafenib in combination with zoledronic acid

CONTACTS AND LOCATIONS:
Locations (1):
- Liver Cancer Institute, Shanghai, Shanghai Municipality, China